CLINICAL TRIAL: NCT04144140
Title: An Open-Label, Multicenter Phase 1/1b Study of Intratumorally Administered STING Agonist E7766 in Subjects With Advanced Solid Tumors or Lymphomas - INSTAL-101
Brief Title: Study of Intratumorally Administered Stimulator of Interferon Genes (STING) Agonist E7766 in Participants With Advanced Solid Tumors or Lymphomas - INSTAL-101
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated earlier due to a business decision; which was unrelated to safety. In addition, there was no clinical activity data that informed the decision.
Sponsor: Eisai Inc. (Industry)
Collaborators: H3 Biomedicine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E7766-G000-101; 2019-000160-17 (EudraCT Number)
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-03

CONDITIONS: Lymphoma; Advanced Solid Tumors
Keywords: Advanced Solid Tumors; E7766; Intratumoral Injection; Stimulator of Interferon Genes Agonist; Interferons; Antineoplastic Agents; Lymphoma; Melanoma; Breast Cancer; Colorectal Cancer; Squamous Cell Carcinoma of the Head and Neck; Oesophageal Squamous Cell Carcinoma; Adenocarcinoma of the Gastroesophageal Junction or Gastric
MeSH Terms: conditions — Lymphoma; Melanoma; Breast Neoplasms; Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation: Advanced Solid Tumors or Lymphomas (Experimental)
  Interventions: Drug: E7766
- Dose Expansion: Advanced Solid Tumors or Lymphomas (Experimental): Dose identified from dose escalation part for E7766 will be used in dose expansion part.
  Interventions: Drug: E7766

INTERVENTIONS:
Drug: E7766 — E7766, solution, intratumorally

SUMMARY:
This is an open label, multicenter, phase 1/1b study to assess safety/tolerability and preliminary clinical activity of E7766 as a single agent administered intratumorally in participants with advanced solid tumors or lymphomas.

DETAILED DESCRIPTION:
The Phase 1/1b study consist of two parts: Dose Escalation and Dose Expansion. In the Dose Escalation Part, E7766 will be administered intratumorally in participants with advanced solid tumors or lymphomas to assess safety/tolerability profile of E7766 and to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of E7766. In the Dose Expansion Part, E7766 at RP2D will be administered to participants with melanoma, head and neck squamous cell carcinoma (HNSCC), breast cancer, colorectal cancer, and/or other tumors including lymphomas to confirm safety and assess preliminary clinical activity of E7766 as a single agent. Clinical activity will be evaluated by objective response rate (ORR), duration of response (DOR), and disease control rate (DCR) on treatment with E7766.

ELIGIBILITY:
1. Participants with solid tumors or lymphomas, confirmed by available histopathology records or current biopsy, that are advanced, nonresectable, or recurrent and progressing since last antitumor therapy, and for which no alternative standard therapy exists.
2. Participants must have a minimum of one injectable lesion which is also accessible for biopsy, and if available, one other measurable lesion also accessible for biopsy.

   An injectable lesion is defined as being measurable (defined below) with a maximum of 3.0 centimeter (cm) longest diameter, accessible for injection as judged by the investigator, and has not been subjected to any prior intratumoral treatment or radiotherapy. Lesions selected for injection must not be too close to a major vessel and not be associated with increased risk of bleeding, example, subcapsular liver lesions or hypervascular tumors.

   Measurable lesions are:
   1. Solid tumors: At least 1 lesion of greater than or equal to (>=1) cm by longest axial diameter or >=1.5 cm short axis diameter if a nodal lesion, which is serially measurable according to modified Response evaluation criteria in solid tumors (RECIST) 1.1 using CT/MRI or photography. Lesions that have had external beam radiotherapy or locoregional therapies such as radiofrequency (RF) ablation must show evidence of progression to be deemed a target lesion.
   2. Lymphoma: At least 1 lymph node with a longest diameter greater than (>)1.5 cm or an extranodal lesion with a longest diameter >1.0 cm
3. Participants with prior Hepatitis B or C are eligible if they have adequate liver function
4. Adequate bone marrow function:

   1. Absolute neutrophil count (ANC) >=1000 per cubic millimeter (/mm^3) (>=1.0*10^3 per microliter [/mcL])
   2. Platelets >=75,000/mm^3 (>=75*10^ 9 per liter [/L])
   3. Hemoglobin >=9.0 grams per deciliter (g/dL)
5. Adequate liver function defined by:

   1. Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) less than or equal to (<=)1.5
   2. Total bilirubin <=1.5*upper limit of the normal range (ULN) except for unconjugated hyperbilirubinemia or Gilbert's syndrome
   3. Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <=3*ULN (in the case of liver metastasis <=5*ULN) unless there are bone metastases. Participants with ALP values >3*ULN and known to have bone metastases can be included.

Exclusion Criteria:

1. Other malignancy active within the previous 2 years except for basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast that has completed curative therapy.
2. Known human immunodeficiency virus (HIV) infection.
3. Major surgery within 4 weeks before the first dose of study drug.
4. Brain metastases that are untreated or in the posterior fossa or involve the meninges. Participants with stable or progressing brain metastases (except in the posterior fossa or involving the meninges) previously treated with brain stereotactic radiotherapy (SRT), whole-brain radiotherapy (WBRT) and/or surgery are allowed as long as the participant is asymptomatic neurologically and does not require immediate local intervention (radiotherapy and/or surgery). In addition, participants must be off immunosuppressive doses of systemic steroids (>10 milligram per day (mg/d) prednisone or equivalent) for at least 4 weeks before study drug administration.
5. Prolongation of corrected QT (QTc) interval to >450 millisecond (msec) for males and females when electrolytes balance is normal.
6. Females who are breastfeeding or pregnant at screening or baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 units per liter (IU/L) or equivalent units of ß-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
7. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (total abstinence [if it is their preferred and usual lifestyle], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 180 days after study drug discontinuation. For sites outside of the European Union, it is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, then the participant must agree to use a medically acceptable method of contraception, that is, double barrier methods of contraception such as condom plus diaphragm or cervical/vault cap with spermicide. If currently abstinent, the participant must agree to use a highly effective method as described above if she becomes sexually active during the study period or for 180 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 28 days before dosing and must continue to use the same contraceptive during the study and for 180 days after study drug discontinuation.
8. Male participants who are partners of women of childbearing potential must use a condom and spermicide and their female partners if of childbearing potential must use a highly effective method of contraception beginning at least 1 menstrual cycle prior to starting study drug(s), throughout the entire study period, and for 180 days after the last dose of study drug, unless the male participants are totally sexually abstinent or have undergone a successful vasectomy with confirmed azoospermia or unless the female partners have been sterilized surgically or are otherwise proven sterile. No sperm donation is allowed during the study period or for 180 days after study drug discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (6):
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Miami Hospital Sylvester Comprehensive Cancer Center, Miami, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pittsburgh Medical Center and Hillman Cancer Center, Pittsburgh, Pennsylvania
- Institut Gustave Roussy, Villejuif, France
- Samsung Medical Center, Seoul, South Korea
- Spain (4):
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid, Madrid
  - INCLIVA Hospital Clínico Universitario de Valencia, Valencia
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United States, France, and United Kingdom from 24 February 2020 to 26 July 2022.
Pre-assignment Details: A total of 31 participants were screened, of which 7 were screen failures and 24 were enrolled to receive study treatment in the Dose Escalation Part of this study. The study was terminated due to sponsor's strategic decision, which is unrelated to safety, therefore no participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part of this study.
Groups:
- Dose Escalation Part: E7766 75 mcg: Participants received E7766 75 microgram (mcg), injection, intratumorally on Days 1, 8, and 15 in the first cycle of 21 days and then on Day 1 of each subsequent 21-days cycle, once every 3 weeks until progressive disease (PD) or until other discontinuation criteria whichever occurred first.
- Dose Escalation Part: E7766 150 mcg: Participants received E7766 150 mcg injection, intratumorally on Days 1, 8, and 15 in the first cycle of 21 days and then on Day 1 of each subsequent 21-days cycle, once every 3 weeks until PD or until other discontinuation criteria whichever occurred first.
- Dose Escalation Part: E7766 300 mcg: Participants received E7766 300 mcg injection, intratumorally on Days 1, 8, and 15 in the first cycle of 21 days and then on Day 1 of each subsequent 21-days cycle, once every 3 weeks until PD or until other discontinuation criteria whichever occurred first.
- Dose Escalation Part: E7766 600 mcg: Participants received E7766 600 mcg injection, intratumorally on Days 1, 8, and 15 in the first cycle of 21 days and then on Day 1 of each subsequent 21-days cycle, once every 3 weeks until PD or until other discontinuation criteria whichever occurred first.
- Dose Escalation Part: E7766 780 mcg: Participants received E7766 780 mcg injection, intratumorally on Days 1, 8, and 15 in the first cycle of 21 days and then on Day 1 of each subsequent 21-days cycle, once every 3 weeks until PD or until other discontinuation criteria whichever occurred first.
- Dose Escalation Part: E7766 1000 mcg: Participants received E7766 1000 mcg injection, intratumorally on Days 1, 8, and 15 in the first cycle of 21 days and then on Day 1 of each subsequent 21-days cycle, once every 3 weeks until PD or until other discontinuation criteria whichever occurred first.
- Dose Expansion Part: Participants were planned to receive the dose identified from dose escalation part for E7766 in dose expansion part. Since no participants were enrolled in the Dose Expansion part of E7766. Hence, no data collection and analysis were done during Dose Expansion part of this study.
Period: Overall Study
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Started | 2 | 2 | 2 | 11 | 6 | 1 | 0
Completed | 2 | 2 | 2 | 11 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received at least 1 dose of study drug. No participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part of this study.
Groups:
- Dose Escalation Part: E7766 75 mcg: Participants received E7766 75 mcg, injection, intratumorally on Days 1, 8, and 15 in the first cycle of 21 days and then on Day 1 of each subsequent 21-days cycle, once every 3 weeks until PD or until other discontinuation criteria whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (4.24) | 53.5 (13.44) | 49.5 (12.02) | 57.4 (12.95) | 60.5 (17.39) | 61.0 (NA) — Standard deviation could not be estimated as there is only one participant in this arm. | 58.5 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 4 | 3 | 0 | 10
  Male | 1 | 1 | 1 | 7 | 3 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 10 | 5 | 1 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 2 | 2 | 2 | 10 | 6 | 1 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Part: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were predefined as any of the following toxicities occurring during Cycle 1 and were assessed by the investigator according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version (v) 5.0. as related to E7766. Nonhematologic toxicity greater than or equal to (>=) Grade 3 (NCI CTCAE v. 5.0), except Grade 3 fatigue less than (<) 5 days. Asymptomatic Grade 3 or 4 laboratory abnormalities that were corrected within 72 hours. >=Grade 3 nausea, vomiting, and diarrhea unless lasting greater than (>) 48 hours despite optimal supportive care. Hematologic toxicity: Grade 4 neutropenia for >=5 days, or febrile neutropenia. Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia with hemorrhage. A DLT may have continued treatment at a reduced dose if the DLT had resolved and in the opinion of the investigator the participant was benefiting from treatment. In case of recurrence of the DLT at a lower dose, E7766 treatment was discontinued.
Time Frame: Cycle 1 (Cycle length= 21 days)
Population: The DLT analysis set included all participants in the Dose Escalation part who completed Cycle 1 without incurring certain major protocol deviations (for instance those related to dosing or others identified before database lock) with at least 2 E7766 injections during Cycle 1 and were evaluable for DLT, or participants who experienced DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 0
Participants | 0 | 0 | 0 | 2 | 1 |

2. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) that emerges during treatment (on or after the first dose of study drug up to 90 days after the participant's last dose) or start day of another anticancer therapy, whichever is earlier; or in case participant has initiated new anticancer therapy within 30 days, then AEs occurring for 30 days following the last dose of E7766, having been absent at pretreatment (Baseline) or reemerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Time Frame: From the first dose of the study drug up to 90 days after the last dose (up to 9 months and 14 days)
Population: The safety analysis set included all participants who received at least 1 dose of study drug. No participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Expansion Part: Participants were planned to receive the dose identified from dose escalation part for E7766 in dose expansion part. Since no participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part of this study.
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1 | 0
Participants | 2 | 2 | 2 | 11 | 6 | 1 |

3. Primary Outcome: Dose Expansion Part: Objective Response Rate Based on Modified Response Evaluation Criteria In Solid Tumors (mRECIST) v1.1
Description: ORR was defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) for target and non-target lesions. CR was defined as the disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in the short axis to less than 10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The tumor assessment was done using number of lesions based on modified RECIST 1.1 as per investigator assessment for assessing tumor burden up to 10 target lesions with up to 5 target lesions per organ.
Time Frame: From date of first dose of study drug until confirmed CR or PR (up to 29 months)
Population: The full analysis set included all participants who received at least 1 dose of study drug. No participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part.
Arm/Group | Dose Expansion Part
Number analyzed (Participants) | 0

4. Primary Outcome: Dose Expansion Part: ORR Based on Immune Response Evaluation Criteria in Solid Tumors (iRECIST)
Description: ORR was defined as the percentage of participants whose BOR was iCR or iPR according to iRECIST as per investigator assessment. iCR: immune complete response achieved with disappearance of all target lesions iCPD: immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions iSD: immune stable disease in the absence of iCR or iPD. iUPD: immune unconfirmed progressive disease when iPD is unconfirmed NE: not evaluable.
Time Frame: From date of first dose of study drug until confirmed iCR or iPR (up to 29 months)
Population: as for outcome 3
Arm/Group | Dose Expansion Part
Number analyzed (Participants) | 0

5. Primary Outcome: Dose Expansion Part: Duration of Response (DOR) Based on mRECIST v1.1
Description: DOR was defined as time from the first documented of CR or PR to the date of first documentation of PD based on modified RECIST 1.1 as per investigator assessment or death (whichever occurs first). CR was defined as the disappearance of all target lesions and non-target lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD for target lesion, was defined as a minimum 20% increase and a minimum 5 mm absolute increase in sum of diameters compared to nadir, or PD for non-target lesion(s) or unequivocal new lesion(s). Nadir was defined as lowest measure sum of diameters of target lesions at any time point from baseline onward. The tumor assessment was done using number of lesions based on modified RECIST 1.1 for assessing tumor burden up to 10 target lesions with up to 5 target lesions per organ.
Time Frame: From first documented confirmed CR or PR until first documentation of PD or death (up to 29 months)
Population: as for outcome 3
Arm/Group | Dose Expansion Part
Number analyzed (Participants) | 0

6. Primary Outcome: Dose Expansion Part: DOR Based on iRECIST
Description: DOR: time from date of first observation of response (iPR or iCR) to date of the first observation of progression based on iRECIST 1.1 as per investigator assessment, or date of death, whatever the cause. iCR: immune complete response achieved with disappearance of all target lesions iCPD: immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first documented confirmed iCR or iPR until first documentation of iPD or death (up to 29 months)
Population: as for outcome 3
Arm/Group | Dose Expansion Part
Number analyzed (Participants) | 0

7. Primary Outcome: Dose Expansion Part: Disease Control Rate (DCR) Based on mRECIST v1.1
Description: DCR was defined as the percentage of participants with a best overall response of CR or PR, or stable disease (SD) based on mRECIST 1.1 as per investigator assessment. Best overall response of SD must have been >=5 weeks after randomization. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference the baseline sum of the diameters of target lesions. SD was when a case does not qualify for either PR or PD and was new non-target lesions. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions.
Time Frame: From first dose of study drug until confirmed CR or PR or >=5 weeks after first dose for SD (up to 29 months)
Population: as for outcome 3
Arm/Group | Dose Expansion Part
Number analyzed (Participants) | 0

8. Primary Outcome: Dose Expansion Part: DCR Based on iRECIST
Description: DCR: percentage of participants with a confirmed iCR, iPR, or i-SD (duration of iSD >=5 weeks). DCR was assessed on iRECIST v1.1 as per investigator assessment. iCR: immune complete response achieved with disappearance of all target lesions iCPD: immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions iSD: immune stable disease in the absence of iCR or iPD. iUPD: immune unconfirmed progressive disease when iPD is unconfirmed NE: not evaluable.
Time Frame: From first dose of study drug until confirmed iCR or iPR or >=5 weeks after first dose for iSD (up to 29 months)
Population: as for outcome 3
Arm/Group | Dose Expansion Part
Number analyzed (Participants) | 0

9. Secondary Outcome: Dose Escalation Part: ORR Based on iRECIST
Description: ORR was defined as the percentage of participants whose BOR was iCR or iPR according to iRECIST as per investigator assessment. iCR: immune complete response achieved with disappearance of all target lesions iCPD: immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions iSD: immune stable disease in the absence of iCR or iPD iUPD: immune unconfirmed progressive disease when iPD is unconfirmed NE: not evaluable.
Time Frame: From date of first dose of study drug until confirmed iCR or iPR (up to 6 months and 18 days)
Population: The full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Dose Escalation Part: ORR Based on mRECIST v1.1
Description: ORR was defined as the percentage of participants with a BOR of CR or PR for target and non-target lesions. CR was defined as the disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in the short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The tumor assessment was done using number of lesions based on modified RECIST 1.1 as per investigator assessment for assessing tumor burden up to 10 target lesions with up to 5 target lesions per organ.
Time Frame: From date of first dose of study drug until confirmed CR or PR (up to 6 months and 18 days)
Population: The full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Dose Escalation Part: DOR Based on iRECIST
Description: as for outcome 6
Time Frame: From first documented confirmed iCR or iPR until first documentation of iPD or death (up to 6 months and 18 days)
Population: The full analysis set included all participants who received at least 1 dose of study drug. Here, Overall number of participants analyzed signifies participants who had overall response (OR) (CR or PR) as per Investigator Assessment.
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Dose Escalation Part: DOR Based on mRECIST v1.1
Description: DOR was defined as time from the first documented of CR or PR to the date of first documentation of PD based on modified RECIST 1.1as per investigator assessment or death (whichever occurs first). CR was defined as the disappearance of all target lesions and non-target lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD for target lesion, was defined as a minimum 20% increase and a minimum 5 mm absolute increase in sum of diameters compared to nadir, or PD for non-target lesion(s) or unequivocal new lesion(s). Nadir was defined as lowest measure sum of diameters of target lesions at any time point from baseline onward. The tumor assessment was done using number of lesions based on modified RECIST 1.1 for assessing tumor burden up to 10 target lesions with up to 5 target lesions per organ.
Time Frame: From first documented confirmed CR or PR until first documentation of PD or death (up to 6 months and 18 days)
Population: The full analysis set included all participants who received at least 1 dose of study drug. Here, Overall number of participants analyzed signifies participants who had OR (CR or PR) as per Investigator Assessment.
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Dose Escalation Part: DCR Based on iRECIST
Description: DCR: percentage of participants with a confirmed iCR, iPR, or i-SD (duration of iSD >=5 weeks). DCR was assessed on iRECIST v1.1 as per investigator assessment. iCR: immune complete response achieved with disappearance of all target lesions iCPD: immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions iSD: immune stable disease in the absence of iCR or iPD iUPD: immune unconfirmed progressive disease when iPD is unconfirmed NE: not evaluable.
Time Frame: From first dose of study drug until confirmed iCR or iPR or >=5 weeks after first dose for iSD (up to 6 months and 18 days)
Population: The full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1
percentage of participants | 100.0 | 0.0 | 50.0 | 36.4 | 16.7 | 0.0

14. Secondary Outcome: Dose Escalation Part: DCR Based on mRECIST v1.1
Description: DCR was defined as the percentage of participants with a best overall response of CR or PR, or SD based on mRECIST 1.1 as per investigator assessment. Best overall response of SD must have been >=7 weeks after randomization. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference the baseline sum of the diameters of target lesions. SD was when a case does not qualify for either PR or PD and was new non-target lesions. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions.
Time Frame: From first dose of study drug until confirmed CR or PR or >=5 weeks after first dose for SD (up to 6 months and 18 days)
Population: The full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1
percentage of participants | 100.0 | 0.0 | 50.0 | 36.4 | 16.7 | 0.0

15. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for E7766
Description: Cmax was quantified using liquid chromatography tandem mass spectrometry (LC-MS/MS) methods.
Time Frame: Dose Escalation: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose; Dose Expansion: Cycle 1 Days 1 and 15: predose up to 2 hours postdose (Cycle length=21 days)
Population: The Pharmacokinetic (PK) analysis set included the group of participants who have received at least 1 dose of study drug and have at least 1 evaluable plasma concentration. No participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part. Here number analyzed "n" are the participants who were evaluable for this outcome measure for given timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Dose Expansion Part: Dose identified from dose escalation part for E7766 was planned be used in dose expansion part. Since no participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part of this study.
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1 | 0
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 4.23 (87.4) | 2.77 (7.16) | 2.95 (9.85) | 8.03 (95.8) | 11.3 (30.6) | 9.99 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. |
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 2 | 1 | 11 | 6 | 0 | 0
  Cycle 1 Day 15 | 1.29 (22.7) | 2.23 (58.1) | 4.53 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 2.72 (168) | 9.33 (34.8) |  |

16. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for E7766
Description: Tmax was quantified using validated liquid LC-MS/MS methods.
Time Frame: as for outcome 15
Population: The PK analysis set included the group of participants who have received at least 1 dose of study drug and have at least 1 evaluable plasma concentration. No participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part.Here number analyzed "n" are the participants who were evaluable for this outcome measure for given timepoints.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1 | 0
hours
  Cycle 1 Day 1 | 0.275 [0.25 to 0.3] | 0.31 [0.27 to 0.35] | 0.275 [0.25 to 0.3] | 0.25 [0.2 to 0.52] | 0.25 [0.2 to 0.28] | 0.28 [0.28 to 0.28] |
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 2 | 1 | 11 | 4 | 0 | 0
  Cycle 1 Day 15 | 0.215 [0.18 to 0.25] | 0.385 [0.27 to 0.5] | 0.25 [0.25 to 0.25] | 0.25 [0.17 to 23.4] | 0.21 [0.2 to 0.25] |  |

17. Secondary Outcome: Part: AUC(0-t): Area Under the Plasma Concentration From Time Zero to Last Curve for E7766
Description: AUC was quantified using validated liquid LC-MS/MS methods.
Time Frame: as for outcome 15
Population: The PK analysis set included the group of participants who have received at least 1 dose of study drug and have at least 1 evaluable plasma concentration. No participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part. Here number analyzed "n" are the participants who were evaluable for this outcome measure for given timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter (h*ng/mL)
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1 | 0
hour*nanograms per milliliter (h*ng/mL)
  Cycle 1 Day 1 | 2.71 (114.0) | 3.42 (64.7) | 4.25 (26.6) | 7.7 (35.9) | 8.29 (44.2) | 10.3 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. |
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 2 | 1 | 11 | 4 | 0 | 0
  Cycle 1 Day 15 | 0.536 (17.0) | 1.95 (29.4) | 5.51 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 4.06 (101.0) | 6.89 (76.9) |  |

18. Secondary Outcome: AUC(0-inf): Area Under the Plasma Concentration From Time Zero to Infinity Curve for E7766
Description: AUC(0-inf) was quantified using liquid chromatography tandem mass spectrometry (LC-MS/MS) methods.
Time Frame: as for outcome 15
Population: The PK analysis set included the group of participants who have received at least 1 dose of study drug and have at least 1 evaluable plasma concentration. No participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part. Here overall number analyzed "N" were the participants who were evaluable for the outcome measure and number analyzed "n" are the participants who were evaluable for given timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 0 | 2 | 2 | 9 | 4 | 1 | 0
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 9 | 3 | 1 | 0
  Cycle 1 Day 1 |  | 5.58 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 4.64 (25.1) | 8.07 (38.5) | 8.93 (54.9) | 10.4 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 2 | 1 | 7 | 4 | 0 | 0
  Cycle 1 Day 15 |  | 2.18 (35.4) | 5.79 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 5.16 (83.6) | 7.07 (75.7) |  |

19. Secondary Outcome: t1/2: Terminal Elimination Half-life for E7766
Description: t1/2 was quantified using validated liquid LC-MS/MS methods.
Time Frame: as for outcome 15
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 0 | 2 | 2 | 9 | 4 | 1 | 0
hour
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 9 | 3 | 1 | 0
  Cycle 1 Day 1 |  | 1.56 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 1.07 (4.61) | 1.18 (36.9) | 1.15 (17.5) | 1 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 2 | 1 | 7 | 4 | 0 | 0
  Cycle 1 Day 15 |  | 0.956 (58.1) | 0.917 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 1.34 (66.7) | 0.723 (59.5) |  |

20. Secondary Outcome: Dose Escalation Part: CL/F: Apparent Total Body Clearance for E7766
Description: CL/F was quantified using validated liquid LC-MS/MS methods.
Time Frame: Dose Escalation: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length=21 days)
Population: The PK analysis set included the group of participants who have received at least 1 dose of study drug and have at least 1 evaluable plasma concentration. As planned, this outcome measure was assessed in dose escalation part only. Here overall number analyzed "N" were the participants who were evaluable for the outcome measure and number analyzed "n" are the participants who were evaluable for given timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 0 | 2 | 2 | 9 | 4 | 1
liter per hour (L/h)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 9 | 3 | 1
  Cycle 1 Day 1 |  | 26.9 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 64.6 (25.2) | 74.4 (38.5) | 87.3 (54.8) | 90.3 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants.
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 2 | 1 | 7 | 4 | 0
  Cycle 1 Day 15 |  | 68.7 (35.3) | 51.8 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 116.0 (83.7) | 110.0 (75.9) |

21. Secondary Outcome: Dose Escalation Part: Vd/F: Apparent Volume of Distribution for E7766
Description: Vd/F was quantified using validated liquid LC-MS/MS methods.
Time Frame: Dose Escalation: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length=21 days)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 0 | 2 | 2 | 9 | 4 | 1
liter
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 9 | 3 | 1
  Cycle 1 Day 1 |  | 60.4 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 100.0 (29.5) | 127.0 (65.9) | 145.0 (50.5) | 131.0 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants.
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 2 | 1 | 7 | 4 | 0
  Cycle 1 Day 15 |  | 94.8 (20.0) | 68.6 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 225.0 (80.0) | 115.0 (40.8) |

22. Secondary Outcome: Dose Escalation Part: CLr: Renal Clearance for E7766
Description: CLr was quantified using validated liquid LC-MS/MS methods.
Time Frame: Dose Escalation: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length=21 days)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 1 | 2 | 11 | 6 | 1
Liter per hour (L/h)
  Cycle 1 Day 1 | 0.0218 (76.3) | 0.0119 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 0.0304 (14.0) | 0.0727 (1030.0) | 0.0474 (54.2) | 0.0256 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants.
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 1 | 1 | 11 | 4 | 0
  Cycle 1 Day 15 | 0.0287 (617.0) | 0.243 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 0.164 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 0.412 (320.0) | 0.0742 (72.9) |

23. Secondary Outcome: Dose Escalation Part: Rac (Cmax): Accumulation Ratio Based on Cmax for E7766
Description: Rac (Cmax) was calculated as the ratio of Cmax on Cycle 1 Day 15 divided by Cmax on Cycle 1 Day 1. Accumulation ratio was quantified using validated liquid LC-MS/MS methods.
Time Frame: Dose Escalation: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length=21 days)
Population: The PK analysis set included the group of participants who have received at least 1 dose of study drug and have at least 1 evaluable plasma concentration. As planned, this outcome measure was assessed in dose escalation part only. Here overall number analyzed "N" were the participants who were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 2 | 1 | 11 | 4 | 0
ratio | 0.305 (126.0) | 0.805 (67.4) | 1.43 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 0.339 (117.0) | 0.892 (10.4) |

24. Secondary Outcome: Dose Escalation Part: Rac (AUC0-t): Accumulation Ratio Based on AUC for E7766
Description: Rac (AUC0-t) was calculated as the ratio of AUC(0-t) on Cycle 1 Day 15 divided by AUC(0-t) on Cycle 1 Day 1. Accumulation ratio was quantified using validated liquid LC-MS/MS methods.
Time Frame: Dose Escalation: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length=21 days)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 2 | 1 | 11 | 4 | 0
ratio | 0.198 (149.0) | 0.571 (30.9) | 1.08 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 0.527 (127.0) | 0.907 (17.2) |

25. Secondary Outcome: Dose Escalation Part: Percentage (Fraction) Excreted (fe) in Urine for E7766
Description: fe was defined as fraction of administered drug (E7766) excreted/recovered in urine. fe was quantified using validated liquid LC-MS/MS methods.
Time Frame: Dose Escalation: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length=21 days)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 1 | 2 | 11 | 6 | 1
percentage of dose
  Cycle 1 Day 1 | 0.0786 (340.0) | 0.0412 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 0.0429 (12.2) | 0.0935 (799.0) | 0.0504 (41.8) | 0.0279 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants.
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 1 | 1 | 11 | 4 | 0
  Cycle 1 Day 15 | 0.0205 (874.0) | 0.386 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 0.302 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 0.279 (167.0) | 0.0655 (30.8) |

26. Secondary Outcome: Dose Escalation Part: Percentage (Fraction) Excreted (fe) in Feces for E7766
Description: fe was defined as fraction of administered drug (E7766) excreted/recovered in feces. fe was quantified using validated liquid LC-MS/MS methods.
Time Frame: Dose Escalation: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length=21 days)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
Number analyzed (Participants) | 2 | 1 | 0 | 1 | 2 | 1
percentage of dose
  Cycle 1 Day 1 | 0.759 (390.0) | 0.573 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. |  | 0.0323 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants. | 0.0274 (85.5) | 0.0963 (NA) — Geometric Coefficient of Variation for this arm was not determined due to insufficient number of participants.
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Progression Free Survival (PFS) Based on mRECIST v1.1
Description: PFS was defined as the time from the first study dose date to the date of first documentation of disease progression or death (whichever occurred first) based on mRECIST v1.1 as per investigator assessment. PD was defined as at least a 20% increase in the sum of LD of target and non-target lesions as compared with the smallest sum of LD and the increase of LD was at least 5 mm (including new lesions).
Time Frame: From first dose of study drug until confirmed PD or death up to 6 months 18 days (Dose Escalation Part) and up to 29 months (Dose Expansion Part)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1 | 0
months | NA [NA to NA] — Median and 95% confidence interval (CI) could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. |

28. Secondary Outcome: PFS Based on iRECIST
Description: PFS was defined as the time from the first dose date to the date of iPD or date of death (whichever occurred first) according to iRECIST version 1.1 as per investigator assessment. iCPD: immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 27
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1 | 0
months | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient events. |

29. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from the date of first dose of study drug until date of death from any cause. OS event was defined as deaths no later than data cut off date or date of death of a participant.
Time Frame: as for outcome 27
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1 | 0
months | NA [NA to NA] — Median and full range could not be estimated due to insufficient events. | NA [NA to NA] — Median and full range could not be estimated due to insufficient events. | NA [NA to NA] — Median and full range could not be estimated due to insufficient events. | NA [NA to NA] — Median and full range could not be estimated due to insufficient events. | NA [NA to NA] — Median and full range could not be estimated due to insufficient events. | NA [NA to NA] — Median and full range could not be estimated due to insufficient events. |

30. Secondary Outcome: Percent Change From Baseline in Tumor Size
Description: Percent change from baseline in tumor size was calculated for the first injected lesion based on Investigator Assessment.
Time Frame: Baseline to up to 6 months and 18 days (Dose Escalation Part) and up to 29 months (Dose Expansion Part)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg | Dose Expansion Part
Number analyzed (Participants) | 2 | 2 | 2 | 11 | 6 | 1 | 0
percent change | NA (NA) — Mean and standard deviation could not be estimated due to insufficient events. | NA (NA) — Mean and standard deviation could not be estimated due to insufficient events. | NA (NA) — Mean and standard deviation could not be estimated due to insufficient events. | NA (NA) — Mean and standard deviation could not be estimated due to insufficient events. | NA (NA) — Mean and standard deviation could not be estimated due to insufficient events. | NA (NA) — Mean and standard deviation could not be estimated due to insufficient events. |

ADVERSE EVENTS:
Time Frame: Dose Escalation Part: From the first dose of the study drug up to 90 days after the last dose (up to 9 months and 14 days)
Description: The safety data was collected for Dose Escalation Part of the study only as no participants were enrolled in the Dose Expansion part of E7766. Hence, no data collection and analysis were done during Dose Expansion part of this study.
Arm/Group | Dose Escalation Part: E7766 75 mcg | Dose Escalation Part: E7766 150 mcg | Dose Escalation Part: E7766 300 mcg | Dose Escalation Part: E7766 600 mcg | Dose Escalation Part: E7766 780 mcg | Dose Escalation Part: E7766 1000 mcg
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/2 | 1/2 | 4/11 | 5/6 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 1/2 | 3/11 | 3/6 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 11/11 | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Part: E7766 75 mcg (N=2) | Dose Escalation Part: E7766 150 mcg (N=2) | Dose Escalation Part: E7766 300 mcg (N=2) | Dose Escalation Part: E7766 600 mcg (N=11) | Dose Escalation Part: E7766 780 mcg (N=6) | Dose Escalation Part: E7766 1000 mcg (N=1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Part: E7766 75 mcg (N=2) | Dose Escalation Part: E7766 150 mcg (N=2) | Dose Escalation Part: E7766 300 mcg (N=2) | Dose Escalation Part: E7766 600 mcg (N=11) | Dose Escalation Part: E7766 780 mcg (N=6) | Dose Escalation Part: E7766 1000 mcg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (7) | 6 (13) | 2 (2) | 0 (0)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (3) | 0 (0)
Oesophageal stent stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (5) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (3) | 1 (4) | 9 (27) | 5 (13) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (11) | 5 (11) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (5) | 2 (10) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 1 (10) | 8 (35) | 5 (19) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (3) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 2 (5) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 4 (4) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (4) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated earlier due to corporate strategic decision, which is unrelated to safety. In addition, there is no clinical activity data that informed the decision. Therefore, no participants were enrolled in the Dose Expansion part. Hence, no data collection and analysis were done during Dose Expansion part of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT04144140/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT04144140/SAP_001.pdf